CLINICAL TRIAL: NCT06278077
Title: Evaluation of the Effects of Neurexan® on Short-Term Insomnia, Daytime Performance and Stress Response by Polysomnography (PSG), Electroencephalogram (EEG), Stress Biomarkers and Patient-Reported Outcomes (PROs)
Brief Title: Neurexan - a Clinical Trial in Short-Term Insomnia Patients
Acronym: NEUREXAN SLEEP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biologische Heilmittel Heel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2104; 2024-514391-41-00 (EU CTIS Number)
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Insomnia; Stress Reaction
Keywords: Polysomnography; Electroencephalogram; Sleep Efficiency; Acute Insomnia; Stress dysregulation; Hyperarousal
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fractures, Stress | interventions — neurexan

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, active- and placebo-controlled confirmatory clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All involved personnel at the investigational site, the Sponsor (except production unit) and the CRO (except independent biostatistician for performing the randomization) will be blinded during the trial. The Investigator keeps the sealed treatment code envelopes throughout the course of the trial for the individual patients and must not break the code without a valid reason (e.g., in case of emergency).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurexan (Experimental): Two tablets taken sublingually 3 times daily for a period of 14 consecutive days, at approximately midday, evening and bedtime and not to be taken with meals.
  Interventions: Drug: Neurexan
- Placebo (Placebo Comparator): Two tablets taken sublingually 3 times daily for a period of 14 consecutive days as for Neurexan
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neurexan — The active ingredients are Passiflora incarnata Dil. D2 (0.6 mg / tablet), Avena sativa Dil. D2 (0.6 mg / tablet), Coffea arabica Dil. D12 (0.6 mg/tablet) and Zincum isovalerianicum Dil. D4 (0.6 mg / tablet). Inactive excipients are lactose monohydrate and magnesium stearate.
  Arms: Neurexan
Drug: Placebo — Contains lactose monohydrate, magnesium stearate and looks identical to Neurexan in terms of taste, size, color and labelling.
  Arms: Placebo

SUMMARY:
This clinical study aims to understand the effects of a medication called Neurexan on sleep patterns and stress in people with short-term insomnia. The study involves comparing Neurexan to a placebo - a tablet that looks like Neurexan but lacks active ingredients. The main goal of the study is to determine if Neurexan can enhance sleep efficiency in those with short-term insomnia. Sleep efficiency, which is the proportion of time spent asleep in relation to total time in bed, including attempts to fall asleep, will be assessed through Polysomnography (PSG). PSG examines various sleep characteristics such as brain activity, muscle and heart activity, and breathing.

Participants will take either Neurexan or the placebo for 14 days. Sleep efficiency will be evaluated using PSG before and after the treatment period. Additionally, sleep quality-related factors will be investigated using PSG data, sleep diaries, and participant-completed questionnaires.

The study will also investigate Neurexan's impact on stress levels. This will be assessed using the Cold Pressor Test, which measures stress through having the participant immerse their hand into ice water, and measuring changes in blood pressure and heart rate, both indicators of stress. In addition, blood and saliva samples collected before and after treatment with Neurexan or placebo, will be analyzed for stress-related hormones such as cortisol. Patient questionnaires and Electroencephalography (EEG), a non-invasive brain activity recording, will further assess stress symptoms.

Researchers will analyze data related to sleep efficiency, sleep quality, and stress symptoms. By comparing outcomes before and after Neurexan or placebo treatment, the study aims to detect improvements in these areas. Positive results with Neurexan but not with the placebo would provide robust evidence for Neurexan's efficacy in addressing sleep and stress management issues. This study contributes valuable insights into Neurexan's potential benefits for individuals with short-term insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Insomnia definition according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria; episode duration less than 3 months.
2. Short-term insomnia with moderate symptoms according to Insomnia Severity Index (ISI) of at least 8 and below 22 being present for at least one week, but no longer than 3 months prior to Screening Visit.
3. Reports habitual bedtime, defined as the time the participant attempts to sleep, between 21:00 and 01:00.
4. Reports regular time spent in bed, either sleeping or trying to sleep, between 6 and 9 hours.
5. ≥18 years of age, not older than 65 years.
6. Legally competent male or female patient.
7. Signed Informed Consent.
8. Females of childbearing potential must agree to maintain highly effective or acceptable birth control throughout the trial (CTFG 2020).
9. Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 at Screening Visit.
10. Use of digital device e.g., smartphone, tablet or laptop.
11. German speaking and reading.

Exclusion Criteria:

1. Patients with insomnia symptoms present longer than 90 days prior to Screening Visit.
2. Based on the diagnostic interview, reported history (within 2 years) of other sleep disorders (e.g., chronic insomnia, circadian rhythm sleep disorders, restless legs syndrome (RLS), obstructive sleep apnea (OSA)), i.e., STOPBang (SBQ) questionnaire score ≥5, International Restless Legs Scale score ≥16).
3. Based on the first polysomnographic screening night at Baseline 1, insomnia due to sleep apnea or periodic limb movement disorder (PLMD): OSA (Apnea Hypopnea Index of >5 events/ hour), PLMD (Periodic Limb Movement Index (PLMI) >15 events/ hour).
4. Rotating shift work with overnight shifts.
5. History of psychiatric disorders within the last 6 months prior to Screening Visit according to the Structured Clinical Interview for DSM-5® Disorders - Clinician Version (SCID-5-CV).
6. History of sensitivity to any component of Neurexan®.
7. Unwilling or unable to comply with all the requirements of the clinical trial protocol.
8. Cognitive impairment (cut-off of 24 points in the Montreal Cognitive Assessment [MoCA]; at Screening Visit.
9. Any history of or current abuse of alcohol and/or amphetamines, benzodiazepines, cocaine, marijuana, methaqualone, methadone, opioids, propoxyphene, barbiturates, phencyclidine; or expected to take during trial participation (urine drug screening at Screening Visit and adaptation nights).
10. Current use of medication affecting sleep, i.e., antidepressants, antipsychotics, diuretics, blood pressure drugs, anti-dementia drugs (e.g., piracetam), herbal and homeopathic medicine, hormone preparations (e.g., thyroxine) with the exception of hormonal contraceptives.
11. Use of Neurexan® within the last two weeks from Screening Visit.
12. Non-pharmacological insomnia therapies (e.g., cognitive behavioral therapy within the last 6 months of Screening Visit, sleep restriction therapy, complementary and alternative therapies as meditation, Traditional Chinese Medicine, aromatherapy).
13. Excessive consumption of xanthine-containing beverages (more than 7 cups daily of coffee or tea or other beverages containing xanthines).
14. Use of nicotine during the last 6 months prior to Screening Visit.
15. Participation in any interventional clinical study within the past 30 days prior to Screening Visit.
16. Any relationship of dependence with the Sponsor or with the Investigator.
17. Active infection/ disease (C-Reactive Protein [CRP] >5 mg/l).
18. Hypertension defined as systolic blood pressure ≥140 mmHg.
19. History of neurological, rheumatic, chronic pain, immune, cardiovascular, pulmonary, liver/ kidney, or metabolic disorder within the last 6 months prior to Screening Visit.
20. Nocturia.
21. Pregnancy (as proven by positive urine pregnancy test at Screening Visit) or breastfeeding.
22. Patients with moderate to severe skin allergies and/or eczema.
23. Raynaud's disease.
24. Donation of blood or platelets 3 months prior to or in-between in-hospital visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Sleep Efficiency. | 14 days
  Sleep Efficiency (SE) assessed using Polysomnography (PSG) is calculated as the ratio of total sleep time to time in bed (i.e., both sleeping and attempting to fall asleep or fall back asleep). SE will be assessed at baseline prior to treatment with investigational drug, then again 14 days later following investigational drug treatment.

SECONDARY OUTCOMES:
Change from baseline in sleep pattern characterized by Number of Awakenings. | 14 days
  Sleep pattern characterized by Number of Awakenings (NWAK) will be assessed using Polysomnography (PSG) at baseline prior to treatment with investigational drug, then again 14 days later following investigational drug treatment.
Change from baseline in daytime performance assessed by Epworth Sleepiness Scale patient questionnaire. | 14 days
  The Epworth Sleepiness Scale (ESS) is a validated measure of a patient's general level of daytime sleepiness. The patient rates their tendency to become sleepy in 8 different situations commonly encountered in daily life, on a scale of 0 (no chance of dozing) to 3 (high chance of dozing). The total ESS score is the sum of each of the 8 scores, with a total score of 0 to 24. The higher the score, the higher the patient's level of daytime sleepiness. A number in the 0-9 range is considered to be normal, whereas a number in the range of 10-24 indicates that expert medical advice should be sought. The ESS will be completed electronically at baseline prior to treatment with investigational drug, then again 14 days later following investigational drug treatment.
Ecological Momentary Assessments - continuous daily stress assessment. | 36 to 56 days
  Patients' perceived stress levels (Ecological Momentary Assessments - EMAs) will be reported electronically at the Screening Visit prior to randomization and treatment with investigational drug, then daily throughout the trial until the Day 28 Follow-up Visit. The questionnaire records levels of stress on a scale of 0 (Not stressed at all) to 10 (Very stressed), as well as the severity of stress (0 - Not severe to 10 - Very severe), how well the patient is managing the stress (0 - Not well to 10 - Very well) and the cause(s) of the stress. No sum score will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Jena University Hospital, Department of Psychiatry & Psychotherapy, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Doering BK, Wegner A, Hadamitzky M, Engler H, Rief W, Schedlowski M. Effects of Neurexan (R) in an experimental acute stress setting--An explorative double-blind study in healthy volunteers. Life Sci. 2016 Feb 1;146:139-47. doi: 10.1016/j.lfs.2015.12.058. Epub 2016 Jan 7. PMID 26772822
- [Background] Herrmann L, Vicheva P, Kasties V, Danyeli LV, Szycik GR, Denzel D, Fan Y, Meer JV, Vester JC, Eskoetter H, Schultz M, Walter M. fMRI Revealed Reduced Amygdala Activation after Nx4 in Mildly to Moderately Stressed Healthy Volunteers in a Randomized, Placebo-Controlled, Cross-Over Trial. Sci Rep. 2020 Mar 2;10(1):3802. doi: 10.1038/s41598-020-60392-w. PMID 32123197
- [Background] Waldschutz R, Klein P. The homeopathic preparation Neurexan vs. valerian for the treatment of insomnia: an observational study. ScientificWorldJournal. 2008 Apr 20;8:411-20. doi: 10.1100/tsw.2008.61. PMID 18454251
- [Background] Dimpfel, W. Effects of Neurexan on Stress-Induced Changes of Spectral EEG Power: A Double-Blind, Randomized, Placebo-Controlled, Crossover Exploratory Trial in Human Volunteers. World Journal of Neuroscience. 2019; 9(3): 100-112.

DOCUMENTS (1):
  • Study Protocol (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT06278077/Prot_000.pdf